CLINICAL TRIAL: NCT05755061
Title: Long-Term Aerobic Walking Exercise for Restoring Cognition and Brain in People With Multiple Sclerosis
Brief Title: WEBCAMS: Walking Exercise for Brain and Cognition in Adults With Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Brian Sandroff, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1194-22
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Relapsing-remitting Multiple Sclerosis
Keywords: Exercise; Cognition; Brain; Rehabilitation; Remote
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEMS Plus (Experimental): Home-based aerobic walking exercise that exceeds published physical activity guidelines for adults with MS
  Interventions: Behavioral: GEMS Plus
- GEMS (Active Comparator): Home-based aerobic walking exercise that meets published physical activity guidelines for adults with MS
  Interventions: Behavioral: GEMS

INTERVENTIONS:
Behavioral: GEMS Plus — 12-months of home-based walking exercise that occurs 3-5 days per week. The program will progress up to intensities that exceed the published physical activity guidelines for adults with MS
  Arms: GEMS Plus
Behavioral: GEMS — 12-months of home-based walking exercise that occurs 3-5 days per week. The program will progress up to intensities that meet the published physical activity guidelines for adults with MS
  Arms: GEMS

SUMMARY:
This study is a randomized controlled trial (RCT) that compares the effects of two different 12-month aerobic walking exercise programs on cognitive processing speed (CPS), brain MRI, and other functional outcomes in 32 adults with multiple sclerosis (MS) who are able to walk without an assistive device but demonstrate slowed CPS. Participants (N=32) will initially undergo screening via telephone, and after satisfying relevant inclusion/exclusion criteria, will provide informed consent, followed by a baseline assessment of CPS remotely via a HIPAA-compliant virtual platform (i.e., Zoom for Healthcare). This assessment will also serve as a screen for ensuring impaired CPS. Following this virtual session, participants will come into Kessler Foundation (KF) and complete a 3-hour baseline assessment (T0) that includes a relatively short battery of neuropsychological tests, a 40-minute MRI scan, tests of walking function, a short questionnaire packet, followed by cardiopulmonary exercise testing on a motor-driven treadmill. Following T0, participants will be randomly assigned into one of the two aerobic walking ET programs that are remotely-delivered and supported by KF research assistants. As the conditions are delivered and supported remotely by KF personnel, the exercise itself takes place in the home/community setting. Both conditions involve behavior coaching via Zoom for Healthcare. The experimental condition involves high-frequency, high-intensity aerobic walking ET that exceeds the published guidelines for physical activity for adults with MS (GEMS+). GEMS + initially involves 10 minutes of moderate intensity aerobic walking exercise for 3 days per week and progresses to upwards of 40 minutes of vigorous intensity aerobic walking exercise for 5 days per week by month 12. The comparison condition involves mild-to-moderate aerobic walking exercise training that approximates published guidelines (GEMS). GEMS initially involves 10 minutes of light intensity aerobic walking exercise for 2 days per week and progresses up to 30 minutes of moderate intensity aerobic walking exercise for 3 days per week. Both conditions further will be monitored based on Fitbit-measured steps per exercise session. Of note, the sample size will be enrolled using 2 overlapping waves (Wave 1 = 14 participants, Wave 2 = 18 participants), 3 months apart. Participants will return to KF at the mid-point (i.e., T6) and end-point (i.e., T12) of the 12-month intervention period to complete the same assessments as T0. The T6 and T12 outcomes will be administered by treatment-blinded research assistants.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis
* Relapse-free for at least 30 days
* Have Internet access on a device larger than a smartphone
* Willingness and ability to travel to Kessler Foundation 3 times over a 12-month period
* Be insufficiently physically active
* Demonstrate low fall risk based on Activities Specific Balance Confidence scores
* Demonstrate low contraindications for exercise
* Right handedness
* English as a primary language
* Demonstrate low cognitive processing speed based on a Zoom-administered Symbol Digit Modalities Test

Exclusion Criteria:

* Acutely taken corticosteroids within 30 days of enrollment
* Use an assistive device (i.e., cane, crutch, walker, rollator) for ambulation
* Experienced a fall in the past 6 months
* Have uncontrolled major depressive disorder or history of bipolar disorder or schizophrenia
* Regularly taking medications that can affect cognition (e.g., antipsychotics, benzodiazepines)
* Demonstrate contraindications for 3T MRI (i.e., having metal/shrapnel in the body, non-MRI compatible aneurysm clips)
* Have severe cognitive impairment causing an inability to follow directions

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive processing speed | Baseline; 6-months; 12-months
  Participants will undertake the Symbol Digit Modalities Test as a cognitive test of cognitive processing speed as one of the primary study outcomes
Change in resting-state functional connectivity | Baseline; 6-months; 12-months
  Participants will undertake an fMRI scan to measure resting-state functional connectivity between the thalamus and other brain regions as one of the primary study outcomes

SECONDARY OUTCOMES:
Change in thalamic volume | Baseline; 6-months; 12-months
  Participants will undertake an MRI scan to measure volume of the thalamus as a secondary study outcome

OTHER OUTCOMES:
Change in aerobic fitness | Baseline; 6-months; 12-months
  Participants will undertake a maximal, graded exercise test on a treadmill to measure aerobic fitness

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided